CLINICAL TRIAL: NCT06088056
Title: A Phase II Study of T-DXd Plus Stereotactic Radiotherapy(SRT) in HER2-positive Breast Cancer Brain Metastases
Brief Title: A Phase II Study of T-DXd Plus SRT in HER2-positive Breast Cancer Brain Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoli Yu, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-BC021
Record Dates: First submitted 2023-07-30; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Brain Metastases; Radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination use of SRT with T-DXd (Experimental): Radiation therapy SRT will be implemented according to investigator's clinical practice(based on brain metastases number and tumor volume). T-DXd(5.4mg/kg, once per 21 days, initiated within 2 weeks after SRT) will be provided to patients with confirmed HER2 positive breast cancer and brain metastasis until tumor progression, a severe adverse event deemed related to the study drug, or death. All dose adjustments should be based on the most severe toxicity level (CTCAE version 5.0) that occurred. Two doses are allowed to be reduced.
  Dose Level 0: 5.4mg/kg Dose Level 1 :4.4mg/kg Dose Level 2: 3.2mg/kg
  Interventions: Drug: Combination use of SRT with T-DXd

INTERVENTIONS:
Drug: Combination use of SRT with T-DXd — Radiation therapy SRT will be implemented according to investigator's clinical practice(based on brain metastases number and tumor volume). T-DXd(5.4mg/kg, once per 21 days, initiated within 2 weeks after SRT) will be provided to patients with confirmed HER2 positive breast cancer and brain metastasis until tumor progression, a severe adverse event deemed related to the study drug, or death. All dose adjustments should be based on the most severe toxicity level (CTCAE version 5.0) that occurred. Two doses are allowed to be reduced.
  Dose Level 0: 5.4mg/kg Dose Level 1 :4.4mg/kg Dose Level 2: 3.2mg/kg

SUMMARY:
This research study will evaluate the efficacy and safety of stereotactic radiotherapy (SRT) combined with Trastuzumab-Deruxtecan (T-DXd; DS-8201a) in HER2-positive Breast Cancer Patients with newly diagnosed or progressing Brain Metastases.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed HER2 positive advanced breast cancer
* Age>18 years.
* Brain metastases confirmed by enhanced brain MRI. Metastases number less than 15.
* KPS≥70 or KPS ≥60 with neurologic symptoms caused by BM
* Life expectancy of more than 6 months
* Prior therapy of oral dexamethasone not exceeding 16mg/d
* Time interval from prior therapy was more than 2 weeks, and evaluation of adverse events is no more than grade 1.
* Screening laboratory values must meet the following criteria( and should be obtained within 28 days prior to registration):

  1. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L, Platelets≥ 90 x 109/L, Hemoglobin ≥ 90 g/L
  2. Aspartate aminotransferase/alanine aminotransferase (AST/ALT) ≤2.5 x ULN without liver metastasis,≤ 5 x ULN with liver metastases
  3. Serum BUN and creatinine ≤ 1.5 x Upper Limit of Normal (ULN)
  4. LVEF ≥ 50%
  5. QTcF < 480 ms
  6. INR≤1.5×ULN，APTT≤1.5×ULN
* Signed the informed consent form prior to patient entry

Exclusion Criteria:

* Leptomeningeal or hemorrhagic metastases
* Uncontrolled epilepsy
* Severe or uncontrolled disease: severe cardiovascular disease, end-stage renal disease, severe hepatic disease, history of immunodeficiency, including HIV positive, active HBV/HCV or other acquired congenital immunodeficiency disease, or organ transplantation history, active infection, etc.
* History of allergy to treatment regimens
* Pregnancy or lactation period， women of child-bearing age who are unwilling to accept contraceptive measures.
* Inability to complete enhanced MRI
* Not suitable for inclusion for specific reasons judged by sponsor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Intracranial objective response rate(IC-ORR) | 2 years
  Proportion of participants with a complete response (CR) or partial response (PR) for intracranial tumors as defined by response assessment in neuro-oncology brain metastases (RANO-BM) criteria.

SECONDARY OUTCOMES:
Intracranial CNS Progression Free Survival(IC-PFS) | 2 years
  Time from treatment until the first date of intracranial disease progression or death due any cause. For participants whose disease has not progressed at the time of the analysis, censoring will be performed using the date of the last valid disease assessment.
Progression Free Survival(PFS) | 2 years
  Time from treatment until the first date of intracranial or extracranial disease progression or death due any cause. For participants whose disease has not progressed at the time of the analysis, censoring will be performed using the date of the last valid disease assessment.
Overall survival(OS) | 3 years
  Time from the treatment until to the date of death, regardless of the cause of death
Percentage of Participants With Adverse Events Percentage of Participants With Adverse Events | 2 years
  Treatment-related adverse events were assessed and graded according to CTCAE v. 5.0
Health-related quality of life per FACT-BR | 2 years
  Health-related quality of life was evaluated using the QLQ-C30 questionnaires to assess Health-related quality of life was evaluated using the FACT-BR questionnaires to assess the quality of life
Local control rate | 2 years
  The percentage of participants who have achieved complete response, partial response and stable disease according to RANO-BM criteria after treatment
Neurocognitive function per HVLT-R | 2 years
  Neurocognitive function was evaluated using HVLT-R test

CONTACTS AND LOCATIONS:
Overall Officials: Zhaozhi Yang, Principal Investigator — Fudan University; Jiayi Chen, Principal Investigator — Ruijin Hospital affiliated to Shanghai Jiaotong University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No